CLINICAL TRIAL: NCT01925066
Title: Optimal Two-Stage Phase 2 Study of Efficacy and Pharmacokinetics of Aerosolized Vancomycin in Methicillin-Resistant Staphylococcus Aureus Pneumonia Under Mechanical Ventilation
Brief Title: Aerosolized Vancomycin in Methicillin-Resistant Staphylococcus Aureus Pneumonia Under Mechanical Ventilation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1206-156-004
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Pneumonia, Staphylococcal; Methicillin-Resistant Staphylococcus Aureus
MeSH Terms: conditions — Pneumonia, Staphylococcal | interventions — Vancomycin; BID protein, human; Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aerosolized Vancomycin (Experimental)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin
  Other Names: 250mg bid, Inhalation for 5-7 days

SUMMARY:
The purpose of this study is to determine whether aerosolized vancomycin is effective in the treatment of methicillin-resistant staphylococcus aureus pneumonia under mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Nosocomial or severe community-acquired pneumonia due to Methicillin-Resistant Staphylococcus aureus
* Must be mechanically ventilated in intensive care unit

Exclusion Criteria:

* Non-bacterial pneumonia, such as viral, fungal, tuberculosis infections
* Underlying respiratory condition: bronchiectasis, post-tuberculosis, chronic obstructive pulmonary disease or asthma
* Complicated pneumonia, such as empyema, parapneumonic effusion requiring chest tube or drainage
* Already or previous treated with intravenous vancomycin (Not pneumonia)
* Adverse reaction due to inhaled ventolin before treatment of aerosolized vancomycin
* Hypersensitivity of vancomycin or glycopeptide antibiotics
* Positive culture of Enterococcus in respiratory specimen
* Pregnant or Breast-feeding patient
* Immunocompromised hosts: more than 1mg/kg of corticosteroid users for more than 3 months, transplantation recipients, AIDS patients
* Another aerosolized antibiotics within 48 hours of study enrollment
* Not adherent to mechanical ventilation protocol of this study
* Not arterial line monitoring
* Vancomycin minimum inhibitory concentration >= 2㎍/㎖ of cultured Staphylococcus aureus

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
clinical cure rate | within the first 30 days after treatment

SECONDARY OUTCOMES:
the peak level of serum vancomycin level | on 3rd and 5th days after treatment

OTHER OUTCOMES:
microbiological response | within the first 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Derived] Cho JY, Kim HS, Yang HJ, Lee YJ, Park JS, Yoon HI, Kim HB, Yim JJ, Lee JH, Lee CT, Cho YJ. Pilot Study of Aerosolised Plus Intravenous Vancomycin in Mechanically Ventilated Patients with Methicillin-Resistant Staphylococcus Aureus Pneumonia. J Clin Med. 2020 Feb 9;9(2):476. doi: 10.3390/jcm9020476. PMID 32050447
- See also: Optimal Two-Stage Designs For Phase II Clinical Trials — http://linus.nci.nih.gov/brb/samplesize/otsd.html